CLINICAL TRIAL: NCT07076459
Title: A Comparative Pharmacokinetic Study of Single-Dose Administration of HR091506 Tablets From Different Batches in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HR091506-104
Record Dates: First submitted 2025-07-15; First posted 2025-07-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-07

CONDITIONS: Health Volunteer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): Period 1: HR091506 tablet T1 Period 2: HR091506 tablet T2 Period 3: HR091506 tablet R
  Interventions: Drug: HR091506 tablet
- Sequence 2 (Experimental): Period 1: HR091506 tablet T2 Period 2: HR091506 tablet R Period 3: HR091506 tablet T1
  Interventions: Drug: HR091506 tablet
- Sequence 3 (Experimental): Period 1: HR091506 tablet R Period 2: HR091506 tablet T1 Period 3: HR091506 tablet T2
  Interventions: Drug: HR091506 tablet
- Sequence 4 (Experimental): Period 1: HR091506 tablet T2 Period 2: HR091506 tablet T1 Period 3: HR091506 tablet R
  Interventions: Drug: HR091506 tablet
- Sequence 5 (Experimental): Period 1: HR091506 tablet T1 Period 2: HR091506 tablet R Period 3: HR091506 tablet T2
  Interventions: Drug: HR091506 tablet
- Sequence 6 (Experimental): Period 1: HR091506 tablet R Period 2: HR091506 tablet T2 Period 3: HR091506 tablet T1
  Interventions: Drug: HR091506 tablet

INTERVENTIONS:
Drug: HR091506 tablet — In each period under fed conditions, subjects received oral administration of either HR091506 tablet（T1）, HR091506 tablet（T2）, or HR091506 tablet（R）.

SUMMARY:
To evaluate the pharmacokinetic characteristics of HR091506 tablets in different batches in healthy subjects after single administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female between the ages of 18 and 50 years, inclusive.
2. At least 50.0 kg for male subjects, 45.0 kg for female subjects, with a Body Mass Index (BMI) between 19.0-26.0 kg/m2, inclusive (BMI = weight/height2).
3. Prior to screening, during the trial, and for 90 days after the last administration, subjects (including male subjects) must not have plans to conceive and must voluntarily adopt effective contraceptive measures.
4. Subjects who could understand the nature, significance, potential benefits, inconvenience, and potential risks of the study, understand the procedures and methods, be willing to complete the trial strictly following the protocol, and voluntarily sign the informed consent.

Exclusion Criteria:

1. Subjects with history of drug or food allergies.
2. Subjects with a history of diseases related to the circulatory, endocrine, nervous, digestive, respiratory, hematolymphatic, immune, mental, skin, bone, muscle, urogenital, mucosal, and metabolic systems.
3. Use of any medication within 14 days prior to dosing.
4. Subjects who have taken any clinical investigational products or participated in the clinical research of medical devices within 90 days before the trial, or plan to participate in other clinical trials during the study.
5. Subjects who have donated blood or experienced blood loss greater than 300 mL, or have received a blood transfusion or used blood products within 90 days prior to screening.
6. Subjects who take more than 5 cigarettes per day on average within 90 days prior to the study or do not agree to prohibit smoking during the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-07-10 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Cmax: Maximum plasma concentration. Blood samples will be collected. | From 0 hour predose up to 36 hours postdose
AUC0-t: Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration. Blood samples will be collected. | From 0 hour predose up to 36 hours postdose
AUC0-∞: Area under the plasma concentration-time curve from time 0 to infinity. Blood samples will be collected. | From 0 hour predose up to 36 hours postdose
Tmax: Observed time to reach Cmax. Blood samples will be collected. | From 0 hour predose up to 36 hours postdose

SECONDARY OUTCOMES:
Incidence of treatment emergent AEs (TEAEs) | From Signing of Informed Consent Form (ICF) up to Safety Follow Up (Up to Day 24)

CONTACTS AND LOCATIONS:
Locations (1):
- Cangzhou Central Hospital, Cangzhou, Hebei, China

IPD SHARING:
Plan to Share IPD: Undecided